CLINICAL TRIAL: NCT02353416
Title: Effect of a Low Glycemic Index Mediterranean Diet on AGEs. A Randomized Clinical Trial
Brief Title: Effect of Low-Glycemic Index Mediterranean Diet on AGEs
Acronym: Nutri_AGEs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis (Other)
Responsible Party: Principal Investigator, Alberto R Osella, Head. Laboratory of Epidemiology and Biostatistics, Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Nutri_AGEs
Record Dates: First submitted 2015-01-28; First posted 2015-02-02 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2015-01

CONDITIONS: Type 2 Diabetes; Insulin Resistance; Obesity; Cardiovascular Disease
Keywords: Mediterranean Diet; Low-Glycemic Index; AGEs
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance; Obesity; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- INRAM guidelines' diet (Placebo Comparator): Intervention in this arm consists in some general dietary advice about healthy dietary components, serving size and frequency of servings following the Italian official guidelines.
  Interventions: Other: INRAM Guidelines' diet
- Low Glycemic Index Mediterranean Diet (Active Comparator): Intervention in this arm consists in a Low Glycemic Index Mediterranean Diet with indication about type of foods than can be consumed frequently (green foods), sometimes (yellow foods) and never (red foods)
  Interventions: Behavioral: Low Glycemic Index Mediterranean Diet

INTERVENTIONS:
Behavioral: Low Glycemic Index Mediterranean Diet — Prescription of a Low Glycemic Index (less than 50) Mediterranean Diet with no more than 10% of total daily calories coming from saturated fats, high in monounsaturated fatty acids (MUFA) from olive oil and omega-3 polyunsaturated fatty acids (ω3PUFA), from both plant and marine sources
  Arms: Low Glycemic Index Mediterranean Diet
Other: INRAM Guidelines' diet — Prescription of INRAM guidelines' diet
  Arms: INRAM guidelines' diet

SUMMARY:
Advanced glycation end products (AGE) result from a chemical reaction between the carbonyl group of reducing sugar and the nucleophilic NH2 of a free amino acid or a protein; lysine and arginine being the main reactive amino acids on proteins. Following this first step, a molecular rearrangement occurs, rearrangement of Amadori resulting to the formation of Maillard products.

DETAILED DESCRIPTION:
Specialized receptors (RAGE, Galectin 3…) bind AGE. The binding to the receptor causes the formation of free radicals, which have a deleterious effect because they are powerful oxidizing agents, but also play the role of intracellular messenger, altering the cell functions.

This role is especially true at the level of endothelial cells as the attachment of AGE to RAGE receptor causes an increase in vascular permeability. AGE binding to endothelium RAGE and to monocytes-macrophages, led to the production of cytokines, growth factors, to the expression of adhesion molecules, and the production of procoagulant activity. Increased permeability, facilitation of leukocyte migration, the production of reactive oxygen species, cytokines and VEGF suggest that the AGE could be an element of a cascade of reactions responsible for the diabetic angiopathy and vascular damages observed during aging and chronic renal failure. Recently, It's been proposed that balanced diets can limit the deleterious effect of AGE. For these reasons, the interest in preventive approaches complementary or alternative to cholesterol reduction should be one of the main objectives of cardiovascular research in the years to come. Already in the '70s the very low incidence of atherosclerotic diseases in Mediterranean countries (Greece and Southern Italy) and the importance of the "dietary factor" in such protection were noticed. Diets for people in these countries are, among other components, very rich in oleic acid, the main constituent of olive oil, with about 29% of daily caloric intake derived from monounsaturated fatty acids. Aim of this trial is to estimate the effect of a Low Glycemic Index Mediterranean Diet on AGE products.

ELIGIBILITY:
Inclusion Criteria:

* Subject enrolled in the Nutriep cohort assembled in 2005-2007

Exclusion Criteria:

* Not enrolled in the Nutriep cohort
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-02; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Advanced glycation end products levels | Six months
  Blood and skin levels of AGEs

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Misciagna, MD, PhD, Study Director — IRCCS Saverio de Bellis. Laboratorio di Epidemiologia e Biostatistica; Rosa Reddavide, Bsc Sc, Study Chair — IRCCS Saverio de Bellis. Laboratorio di Epidemiologia e Biostatistica
Locations (2):
- Italy (2):
  - Laboratory of Epidemiology and Biostatistics, IRCCS Saverio de Bellis, Castellana Grotte, BA
  - Laboratory of Epidemiology and Biostatistics, Castellana Grotte, BA

REFERENCES:
- [Background] Cozzolongo R, Osella AR, Elba S, Petruzzi J, Buongiorno G, Giannuzzi V, Leone G, Bonfiglio C, Lanzilotta E, Manghisi OG, Leandro G; NUTRIHEP Collaborating Group; Donnaloia R, Fanelli V, Mirizzi F, Parziale L, Crupi G, Detomaso P, Labbate A, Zizzari S, Depalma M, Polignano A, Lopinto D, Daprile G. Epidemiology of HCV infection in the general population: a survey in a southern Italian town. Am J Gastroenterol. 2009 Nov;104(11):2740-6. doi: 10.1038/ajg.2009.428. Epub 2009 Jul 28. PMID 19638964
- [Derived] Hooper L, Abdelhamid AS, Jimoh OF, Bunn D, Skeaff CM. Effects of total fat intake on body fatness in adults. Cochrane Database Syst Rev. 2020 Jun 1;6(6):CD013636. doi: 10.1002/14651858.CD013636. PMID 32476140